CLINICAL TRIAL: NCT07373418
Title: GLOW UP: A Single-Center Observational Study Developing Digital Biomarkers for Prediabetes Screening and Lifestyle Phenotyping
Brief Title: Glucose Observation and Wearable Use for Prevention
Acronym: GlowUp
Status: Recruiting | Type: Observational
Sponsor: University of St.Gallen (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00972
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prevention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prediabetic: Adults aged ≥45 years with BMI ≥25 kg/m².
  FPG 5.6-6.9 mmol/L and/or HbA1c 5.7-6.4% (clinical prediabetes thresholds).
  No known type-2 diabetes diagnosis.
- Normoglycemic: Adults aged ≥45 years with BMI ≥25 kg/m². FPG <5.6 mmol/L and HbA1c <5.7% (normoglycemic; no prediabetes). No known type-2 diabetes diagnosis.

SUMMARY:
The GLOW UP study is a single-center, prospective, observational case-control study conducted in St. Gallen, Switzerland. The primary aim of the study is to examine to what degree lifestyle data collected from wearable devices and a smartphone app can identify individuals with prediabetes (vs. normoglycemic) in a real-world setting. The study also aims to characterize variability in lifestyle and glycemic patterns and to examine how between- and within-person differences relate to diabetes risk; to identify personalized predictors of early metabolic dysregulation. The study also evaluates new image-based meal tracking algorithms for predicting glycemic control and examines how reminder messages influence adherence to a ~4-week meal logging protocol.

The study aims to enroll 200 adults aged 45 years and older with a BMI of at least 25 kg/m² and no known diagnosis of diabetes, including 100 participants with prediabetes and 100 normoglycemic (metabolically healthy) controls. Participants will be classified at the baseline visit using HbA1c and fasting plasma glucose (FPG) tests, with prediabetes defined as HbA1c 5.7-6.4% and/or FPG 5.6-6.9 mmol/L, and normoglycemia defined as HbA1c <5.7% and FPG <5.6 mmol/L, following clinical standards. During the ~4-week observational period, participants will be asked to wear a smart ring, a wrist-worn smartwatch, and a blinded continuous glucose monitor (CGM). Participants will be asked to log/take-images of their meals via a study app and to complete brief questionnaires (e.g., tracking mood, stress, and contextual meal annotations) via ecological momentary assessments. FPG and HbA1c samples will be collected at baseline to classify participants as prediabetic or normoglycemic, and again at follow-up (~4 weeks), which will serve as the primary outcome to evaluate associations between lifestyle and wearable-derived data and diabetes risk status.

ELIGIBILITY:
Inclusion Criteria:

* Citizens or residents of Switzerland who are German-speaking (main place of living or employment in Switzerland).
* Age ≥45 years.
* BMI ≥25 kg/m² (overweight or obese).
* Regular access to a smartphone (iOS or Android) with a data plan.
* Able to use smartphone applications.
* Able to walk independently.

Exclusion Criteria:

* History of stroke, heart disease, renal failure, cancer, or diabetes (type 1 or type 2).
* Past vascular bypass surgery or angioplasty.
* Current or planned use of glucose-lowering medications during the upcoming 4 weeks (e.g., GLP-1 receptor agonists, metformin).
* Pregnant or breastfeeding.
* Relevant skin conditions at wearable placement sites (e.g., upper arm).
* BMI <25 kg/m² confirmed at enrollment.
* FPG ≥7.0 mmol/L and/or HbA1c ≥6.5% (newly identified type 2 diabetes); Individuals who meet type-2 diabetes criteria at enrollment, based on Swiss/ADA diagnostic criteria will be informed of blood test results and referred to a GP. These individuals will be deemed ineligible and excluded from the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults ≥45 years with BMI ≥25 kg/m², German-speaking residents of Switzerland, without known diabetes, recruited from GP practices, community and workplace channels, and general public advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes risk status (prediabetic vs. normoglycemic) | At follow-up, week 4
  Prediabetic (FPG levels 5.6-6.9mmol/L and/or HbA1c levels 5.7%-6.4%) Normoglycemic (FPG levels <5.6mmol/L and HbA1c levels <5.7%)

SECONDARY OUTCOMES:
Diabetes risk at alternative FPG and HbA1c thresholds | At follow-up, week 4
  Participants will also be classified using alternative FPG and HbA1c thresholds based on the observed distribution of glycemic values in the resulting study sample (e.g., high-risk prediabetes FPG ≥6.0 mmol/L, HbA1c ≥6.0%). Additionally, continuous FPG and HbA1c values will be analyzed.
Metabolic phenotypes | At follow-up, week 4
  Metabolic phenotypes defined based on a combination of FPG, HbA1c, body mass index (BMI) and visceral fat levels.
Continuous glycemic control | Up to 4 weeks
  Continuous glucose levels (mmol/L) over the ~4-week period to characterize dynamic glucose patterns.
Lifestyle profiles | Up to 4 weeks
  Lifestyle patterns derived based on nutrition (e.g., macro-nutrient composition), physical activity, sleep, stress levels (e.g., survey-based, HR/HRV).
Adherence to image-based food tracking | Up to 4 weeks
  Number of meal logs completed

CONTACTS AND LOCATIONS:
Locations (1):
- HOCH Health and School of Medicine, University of St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided